CLINICAL TRIAL: NCT06980610
Title: A RANDOMIZEZ OPEN CONTROLLED CLINICAL TRIAL COMPARING THE MEN HEALING TIME WITH COLLATAMP VERSUS DIRECTED HEALING IN DIGESTIVE STOMA CLOSSURES
Brief Title: A Randomized Open Controlled Clinical Trial Comparing the Mean Healing Time With Collatamp Versus Directed Healing in Digestive Stoma Closures
Acronym: CLvsCD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-A02240-47
Record Dates: First submitted 2025-05-19; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Surgery, Colorectal
Keywords: SURGERY,; digestive stoma closures

STUDY DESIGN:
Intervention Model Description: Interventional research with minimal risks and constraints, not involving a product mentioned in Article L. 5311-1 of the CSP
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COLLATAMP (Experimental): The strategy under research is the surgical technique with Collatamp interposition between the musculoaponeurotic plane and the cutaneous plane during stoma closures.
  Interventions: Procedure: digestive stoma closures
- directed healing (Active Comparator): The strategy used as a reference is the surgical technique of directed healing, with the use of an Algosteril wick.
  Interventions: Procedure: digestive stoma closures

INTERVENTIONS:
Procedure: digestive stoma closures — Both surgical techniques (Collatamp interposition and directed healing) are routinely used in the CVMC and Digestive Cancer Surgery departments for stoma closure or restoration of digestive continuity. The choice of technique is at the surgeon's discretion.
  Specific procedures related to the research:
  Procedures that differ from standard management are randomization and patient completion of a questionnaire.

SUMMARY:
The process of directed healing is a slow one, not without any constraints for patients. In contact with the intestinal flora during the stoma time, the tissues harboring digestive bacteria do not allow direct skin closure without the risk of complications during the restoration of digestive continuity after having to perform an ileal or colonic stoma. Collatamp interposition would allow direct wound closure without additional complications. Various studies have compared directed healing and direct skin closure during stoma closure/restoration of continuity. Overall, directed healing reduces the risk of infection, abscesses, and surgical time, but results in greater constraints for the patient, i.e., longer healing time, more pain, and a poorer cosmetic result compared to direct skin closure.

ELIGIBILITY:
Inclusion Criteria:

* Person having received full information on the organization of the research and having signed their informed consent
* Patients aged 18 and over
* Patients requiring ileostomy or colostomy closure, or restoration of digestive continuity
* Person affiliated with a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Patient suffering from an immune deficiency (which would alter the healing process)
* Patient unable to complete the questionnaire
* Patient with a known intolerance, hypersensitivity, or allergy to aminoglycosides or bovine collagen
* Patient suffering from myasthenia gravis
* Woman of childbearing age without effective contraception
* Person referred to in Articles L. 1121-5, L. 1121-7, and L. 1121-8 of the French Public Health Code
* Pregnant woman, woman in labor, or breastfeeding mother
* Minor (non-emancipated)
* Adult subject to a legal protection measure (guardianship, curatorship, or legal protection)
* Adult unable to express consent . Person deprived of liberty by a judicial or administrative decision, person receiving psychiatric care pursuant to Articles L. 3212-1 and L. 3213-1

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Time until complete healing expressed in days | 6 months maximum
  Duration of participation of the person participating in the research (including the follow-up period): 6 months maximum
  Duration of statistical analysis and provision of the final report:
  12 months

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol